CLINICAL TRIAL: NCT04431661
Title: CAOCT Study is a Prospective, Multi-centre, Single Cohort, Diagnostic Accuracy Study, Planned to Include 131 Patients in About 3 European Countries After Successful Return of Spontaneous Circulation After Out of Hospital Cardiac Arrest
Brief Title: CAOCT: Intra CoronAry Optical Computerized Tomography in out-of Hospital Cardiac Arrest Patients
Status: Terminated | Type: Observational
Why Stopped: Low patient recruitment rate and change of hopsital procedures for handling cardiac arrest patients during emergency
Sponsor: Ceric Sàrl (Industry)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: The CAOCT Study
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Out of Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Optical Coherence Tomography — OCT (DragonFly, Abbott Vascular) will be performed after angiography. OCT images will be acquired using the 6F guide catheter compatible DragonFly System (Abbott Vascular, Santa Clara, USA). The catheter will be introduced into the first coronary artery via a standard 0.014-inch angioplasty wire, after prior injection of an intracoronary bolus of nitro-glycerine (according to the hemodynamic conditions of the patient). To remove all blood adequately from the imaging site, nonocclusive flushing will be performed using continuously inject via an automated power injector, and the OCT catheter will be pulled back at a speed of 18 mm/second to guarantee sufficient time to acquire images of a 54 mm long segment (frame density: 10 frames/mm).
Procedure: Coronary Angiography — The coronary angiography will be performed according to the strategies described in the consensus statement from the European Association for Percutaneous Cardiovascular Interventions (EAPCI)/Stent for Life (SFL) groups.Transradial or transfemoral 6F/7F approaches are recommended. The choice of diagnostic catheters, guiding catheters, guidewires, pre-dilatation, atherectomy devices, and post dilatation is let to the investigator's discretion.
Procedure: Per cutaneous coronary intervention — Based on coronary angiography and OCT analyses by the investigators, PCI will be performed, preferentially for the identified culprit lesion(s) only. The guiding catheters, guidewires, pre-dilatation, atherectomy devices, and post dilatation are left to physician discretion. The use of semi- or non-compliant balloons number and diameter of drug eluting stent(s) will also be left to the physician discretion, but post dilation will be strongly recommended in case of PCI. OCT can eventually be performed after stent implantation to guide, post dilation strategy.

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) is a leading cause of sudden death in Europe and the United States. Mortality is currently close to 40% among those patients who had been successfully resuscitated after OHCA associated with ventricular fibrillation or pulseless ventricular tachycardia . Coronary artery disease is observed in up to 70% of patients with OHCA and immediate coronary angiography . Current European and American guidelines recommend immediate coronary angiography with primary angioplasty in OHCA patients with ST-segment elevation on ECG after successful resuscitation . Furthermore, the identification of the culprit lesion by coronary angiography among patients with an acute coronary syndrome (ACS) and no OHCA is challenging. In a recent cardiac magnetic resonance study, Heitner et al. found that in almost half of the patients with non-ST segment elevation ACS, the culprit lesion was not properly detected or identified by coronary angiography. In the Coronary Angiography after cardiac arrest (COACT) trial, a randomized controlled trial comparing immediate versus delayed coronary angiography after OHCA in patients without ST segment elevation on ECG, some degree of coronary artery disease was found in 64.5% of the patients in the immediate angiography group and an unstable coronary lesion was identified in only 13.6% of the patients. However, in survivors of OHCA without ST segment elevation on ECG, the use of intra coronary optical computerized tomography (OCT) led to identification of plaque rupture (27%), plaque erosion (36%) and coronary thrombosis (59%) undetected on angiography. There is hence a clear need to improve causality diagnosis among patients resuscitated after OHCA and without ST segment elevation on ECG, and, in the case of coronary artery disease detection, to better identify the culprit vessel/lesion ultimately leading to a targeted treatment. These are the reasons why we have designed a prospective, multi-centre, single cohort, diagnostic accuracy study: to better explore the incidence of a true ACS among OHCA survivors and to evaluate the accuracy of angiography to detect the culprit lesion when compared to OCT.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of age ≥ 18 years and ≤ 85 years,
* The delay between OHCA and basic life support (no flow period) is ≤ 5 minutes,
* First recorded ECG exhibits a shockable rhythm (ventricular tachycardia/ventricular fibrillation).

Exclusion Criteria:

* The patient is still receiving cardiac massage at the time of admission in the cath-lab,
* There is an obvious extra cardiac cause to the cardiac arrest (suicide, drowning, hanging, trauma etc.),
* The patient has prior coronary artery bypass grafting,
* The patient has incessant ventricular tachycardia/fibrillation,
* The patient has at least one acute or chronic coronary occlusion of an epicardial coronary artery ≥2.0mm of diameter on conventional angiography, The coronary artery anatomy does not allow realization of three vessels OCT according to the interventional cardiologist (severe tortuosity, severe calcifications etc.),
* The patient is in cardiogenic shock or with a left ventricular assistance device,
* The post ROSC ECG (12 leads) exhibits ST segment elevation (defined as a ≥1mm ST segment elevation in two or more contiguous standard leads or as a ≥2mm ST segment elevation in two or more precordial leads),
* The post ROSC ECG (12 leads) exhibits new left bundle block branch (LBBB).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All OHCA patients with no obvious non-cardiovascular reason managed by a pre-hospital emergency system will be screened for inclusion in the study
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of misclassification of at least one unstable coronary artery lesion per patient, between core lab angiography and core lab OCT assessments. | Intra operative, up to 12 months
  The core lab OCT analysis is considered as the gold standard for unstable coronary lesion detection.
  Detection of unstable coronary lesion by OCT includes atherosclerosis plaque rupture/erosion and thrombosis, calcified noduli with apposed thrombus, and spontaneous coronary dissection.
  Angiographically, unstable coronary lesions are defined as coronary lesions with at least >50% stenosis and the presence of characteristics of plaque disruption, including irregularity, dissection, haziness, or thrombus.
  A misclassification is either an unstable lesion detected by core lab OCT and misdiagnosed or undiagnosed on core lab angiography, or an unstable lesion as defined on core lab angiography but without plaque rupture/erosion and thrombosis, calcified noduli with apposed thrombus, and spontaneous coronary dissection on core lab OCT.

SECONDARY OUTCOMES:
The misclassification rate per coronary artery segment analysis, on angiography versus OCT (both techniques peri procedural as assessed by investigators) | Intra operative, up to 12 months
  All analysable coronary segments according to the American Heart Association (AHA) classification (8) will be included in the final analysis. All paired (peri procedural as assessed by investigators angio and OCT) analysed segments will be included in the analysis.
The percentage of patients for whom peri procedural OCT findings change their management (including revascularization strategy) when compared to the initial therapeutic strategy decided upon after investigator-assessed on-line angiography | Intra operative, up to 12 months
  This endpoint represents a comparison between the management of the culprit lesion identified by the investigator after coronary angiography (and strictly captured in the electronic Case Report Form (eCRF) before OCT) and management of the culprit lesion as identified after OCT. Change in interventional management will include patients in whom an initially planned PCI was hold off after OCT and, vice versa, those declined a PCI in whom a PCI was finally decided after OCT. A patient for whom angiography and OCT-based diagnosis would lead to PCI of an additional but distinct coronary segment within the same vessel will be considered as a change in PCI plan.
The percentage of unstable lesions (core lab OCT) intended to be left untreated by PCI after peri procedural (as assessed by investigators) angiography | Intra operative, up to 12 months
  The percentage of unstable lesions as defined by the core lab OCT core lab that were not defined as potential culprit lesion by the investigators after conventional angiography. This will reflect the incidence of undiagnosed and untreated coronary culprit coronary lesion after OHCA.
The percentage of stable lesions (core lab OCT) intended to be treated by PCI after peri procedural (as assessed by investigators) conventional angiography | Intra operative, up to 12 months
  A stable lesion will be defined as a coronary stenosis ≥20% without any features of instability (no plaque rupture or erosion, no thrombosis) on core-lab OCT.
The percentage of misclassification for unstable lesion between peri procedural (as assessed by investigators) OCT and core lab OCT analysis. | Intra operative, up to 12 months
  The unstable lesion as detected during the procedure by the investigator and compared with the corelab analysis.
The duration of the procedure | Intra operative, up to 12 months
  Duration on the procedure will include timing from arterial sheath insertion to final run of angiography (angio), to final run of OCT (intracoronary imaging), and from the end of the angiography or intra coronary imaging to the end of the PCI procedure when applicable (Usually between set puncture to introducer removal).
The irradiation during the procedure | Intra operative, up to 12 months
  Patient irradiation will be determined after conventional angiography (angio), after OCT procedure (intracoronary imaging), and after PCI when applicable (angioplasty). Total procedural irradiation will also be calculated as the cumulative irradiation received during angio, intracoronary imaging and PCI if applicable.
The volume of contrast dye injection | Intra operative, up to 12 months
  The volume of contrast dye injection will be determined after conventional angiography (angio), after OCT procedure (intracoronary imaging), and after PCI when applicable (angioplasty). Total volume of contrast dye injection will also be calculated as the cumulative volume injected during angio, intracoronary imaging and PCI when applicable
The rate of OCT-related complications | Intra operative, up to 12 months
  The OCT related complications include coronary dissection, perforation, plaque embolization etc.
The rate of Major Adverse Coronary and Cerebrovascular Events (MACCE). | Day 1, Day 30 and Day 90
  The MACCE evaluation will include all-cause mortality, myocardial infarction, stroke, ischemia driven target lesion revascularization.
The rate of all-cause mortality | Day 1, Day 30, Day 90 and Day 365
  This includes all cause mortality rate
The rate of stent thrombosis | Day 1, Day 30 and Day 90
  According to Academic Research Consortium-2 (ARC2) definition

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Varenne, MD, PHD, Principal Investigator
Locations (7):
- UZ Leuven, Leuven, Belgium
- France (5):
  - CHU Gabriel-Montpied, Clermont-Ferrand
  - CHU Timone Adultes, Marseille
  - Hôpital Lariboisière, Paris
  - Hôpital Cochin, Paris
  - CHU Toulouse Rangueil, Toulouse
- Clinical Center of Serbia. School of medicine, Belgrade, Serbia

REFERENCES:
- [Background] McDonnell SJ, Gates S, Perkins GD. Utstein recommendations for reporting out of hospital cardiac arrest (OHCA) registry studies-A review of the literature. Resuscitation. 2017;118:e103.
- [Background] Miller LM, Gal A. Cardiovascular system and lymphatic vessels. Pathologic basis of veterinary disease. 2017:561.
- [Background] Hepler MD, Schafer MF. Chapter 18 - Surgical Treatment of Lumbar Spinal Disorders. In: Benzon HT, Rathmell JP, Wu CL, Turk DC, Argoff CE, editors. Raj's Practical Management of Pain (Fourth Edition). Philadelphia: Mosby; 2008. p. 389-400.
- [Background] Marso SP. 23 - Revascularization Approaches. In: de Lemos JA, Omland T, editors. Chronic Coronary Artery Disease: Elsevier; 2018. p. 337-54.
- [Background] Ibrahim K, editor Increased rate of stentthrombosis due to clopidogrel resistance in patients in therapeutic hypothermia after sudden cardiac death. European Heart Journal; 2011: OXFORD UNIV PRESS GREAT CLARENDON ST, OXFORD OX2 6DP, ENGLAND.
- [Result] Degrell P, Picard F, Combaret N, Mogi S, Motreff P, Cariou A, Varenne O. Coronary atherothrombosis in cardiac arrest survivors without ST-segment elevation on ECG. Resuscitation. 2019 Jun;139:189-191. doi: 10.1016/j.resuscitation.2019.01.046. Epub 2019 Mar 27. No abstract available. PMID 30928505
- [Result] Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, Onuma Y, Morel MA, van Es GA, Zuckerman B, Fearon WF, Taggart D, Kappetein AP, Krucoff MW, Vranckx P, Windecker S, Cutlip D, Serruys PW; Academic Research Consortium. Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document. Circulation. 2018 Jun 12;137(24):2635-2650. doi: 10.1161/CIRCULATIONAHA.117.029289. PMID 29891620
- [Result] Heitner JF, Senthilkumar A, Harrison JK, Klem I, Sketch MH Jr, Ivanov A, Hamo C, Van Assche L, White J, Washam J, Patel MR, Bekkers SCAM, Smulders MW, Sacchi TJ, Kim RJ. Identifying the Infarct-Related Artery in Patients With Non-ST-Segment-Elevation Myocardial Infarction. Circ Cardiovasc Interv. 2019 May;12(5):e007305. doi: 10.1161/CIRCINTERVENTIONS.118.007305. PMID 31035776
- [Result] Lemkes JS, Janssens GN, van der Hoeven NW, Jewbali LSD, Dubois EA, Meuwissen M, Rijpstra TA, Bosker HA, Blans MJ, Bleeker GB, Baak R, Vlachojannis GJ, Eikemans BJW, van der Harst P, van der Horst ICC, Voskuil M, van der Heijden JJ, Beishuizen A, Stoel M, Camaro C, van der Hoeven H, Henriques JP, Vlaar APJ, Vink MA, van den Bogaard B, Heestermans TACM, de Ruijter W, Delnoij TSR, Crijns HJGM, Jessurun GAJ, Oemrawsingh PV, Gosselink MTM, Plomp K, Magro M, Elbers PWG, van de Ven PM, Oudemans-van Straaten HM, van Royen N. Coronary Angiography after Cardiac Arrest without ST-Segment Elevation. N Engl J Med. 2019 Apr 11;380(15):1397-1407. doi: 10.1056/NEJMoa1816897. Epub 2019 Mar 18. PMID 30883057
- [Result] Noc M, Fajadet J, Lassen JF, Kala P, MacCarthy P, Olivecrona GK, Windecker S, Spaulding C; European Association for Percutaneous Cardiovascular Interventions (EAPCI); Stent for Life (SFL) Group. Invasive coronary treatment strategies for out-of-hospital cardiac arrest: a consensus statement from the European association for percutaneous cardiovascular interventions (EAPCI)/stent for life (SFL) groups. EuroIntervention. 2014 May;10(1):31-7. doi: 10.4244/EIJV10I1A7. PMID 24832635
- [Result] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; American College of Emergency Physicians; Society for Cardiovascular Angiography and Interventions. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines: developed in collaboration with the American College of Emergency Physicians and Society for Cardiovascular Angiography and Interventions. Catheter Cardiovasc Interv. 2013 Jul 1;82(1):E1-27. doi: 10.1002/ccd.24776. Epub 2013 Jan 8. No abstract available. PMID 23299937
- [Result] Patel N, Patel NJ, Macon CJ, Thakkar B, Desai M, Rengifo-Moreno P, Alfonso CE, Myerburg RJ, Bhatt DL, Cohen MG. Trends and Outcomes of Coronary Angiography and Percutaneous Coronary Intervention After Out-of-Hospital Cardiac Arrest Associated With Ventricular Fibrillation or Pulseless Ventricular Tachycardia. JAMA Cardiol. 2016 Nov 1;1(8):890-899. doi: 10.1001/jamacardio.2016.2860. PMID 27627616
- [Result] Roger VL, Weston SA, Killian JM, Pfeifer EA, Belau PG, Kottke TE, Frye RL, Bailey KR, Jacobsen SJ. Time trends in the prevalence of atherosclerosis: a population-based autopsy study. Am J Med. 2001 Mar;110(4):267-73. doi: 10.1016/s0002-9343(00)00709-9. PMID 11239844
- [Result] Zahger D. Immediate coronary angiography in survivors of out-of-hospital cardiac arrest. N Engl J Med. 1997 Oct 30;337(18):1321-2. doi: 10.1056/NEJM199710303371816. No abstract available. PMID 9380089
- [Result] Spaulding CM, Joly LM, Rosenberg A, Monchi M, Weber SN, Dhainaut JF, Carli P. Immediate coronary angiography in survivors of out-of-hospital cardiac arrest. N Engl J Med. 1997 Jun 5;336(23):1629-33. doi: 10.1056/NEJM199706053362302. PMID 9171064
- [Result] Jiangping S, Zhe Z, Wei W, Yunhu S, Jie H, Hongyue W, Hong Z, Shengshou H. Assessment of coronary artery stenosis by coronary angiography: a head-to-head comparison with pathological coronary artery anatomy. Circ Cardiovasc Interv. 2013 Jun;6(3):262-8. doi: 10.1161/CIRCINTERVENTIONS.112.000205. Epub 2013 May 21. PMID 23696600
- [Result] Penela D, Magaldi M, Fontanals J, Martin V, Regueiro A, Ortiz JT, Bosch X, Sabate M, Heras M. Hypothermia in acute coronary syndrome: brain salvage versus stent thrombosis? J Am Coll Cardiol. 2013 Feb 12;61(6):686-7. doi: 10.1016/j.jacc.2012.10.029. Epub 2012 Dec 19. No abstract available. PMID 23265329
- [Result] Joffre J, Varenne O, Bougouin W, Rosencher J, Mira JP, Cariou A. Stent thrombosis: an increased adverse event after angioplasty following resuscitated cardiac arrest. Resuscitation. 2014 Jun;85(6):769-73. doi: 10.1016/j.resuscitation.2014.02.013. Epub 2014 Feb 23. PMID 24572484
- [Result] Bjelland TW, Hjertner O, Klepstad P, Kaisen K, Dale O, Haugen BO. Antiplatelet effect of clopidogrel is reduced in patients treated with therapeutic hypothermia after cardiac arrest. Resuscitation. 2010 Dec;81(12):1627-31. doi: 10.1016/j.resuscitation.2010.07.002. Epub 2010 Aug 19. PMID 20727659
- [Result] Rosencher J, Gouffran G, Bougouin W, Varenne O. Optimal antiplatelet therapy in out-hospital cardiac arrest patients treated by primary percutaneous coronary intervention. Resuscitation. 2015 May;90:e7-8. doi: 10.1016/j.resuscitation.2015.02.030. Epub 2015 Mar 7. No abstract available. PMID 25758639
- [Result] Adrie C, Adib-Conquy M, Laurent I, Monchi M, Vinsonneau C, Fitting C, Fraisse F, Dinh-Xuan AT, Carli P, Spaulding C, Dhainaut JF, Cavaillon JM. Successful cardiopulmonary resuscitation after cardiac arrest as a "sepsis-like" syndrome. Circulation. 2002 Jul 30;106(5):562-8. doi: 10.1161/01.cir.0000023891.80661.ad. PMID 12147537